CLINICAL TRIAL: NCT05692856
Title: Muscle Memory After Treatment With Anabolic Substance Clenbuterol and Resistance Training in Humans: Myonuclear Addition, Hypertrophy and Myocellular Reprogramming
Brief Title: Muscle Memory After Treatment With Anabolic Substance Clenbuterol and Resistance Training in Humans
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Morten Hostrup, PhD (Other)
Responsible Party: Sponsor-Investigator, Morten Hostrup, PhD, Associate Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CLEN-MEM
Record Dates: First submitted 2022-12-23; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Skeletal Muscle Physiology
MeSH Terms: interventions — Clenbuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clenbuterol (Experimental): Participants are randomized to daily ingestion of clenbuterol for a period of 8 weeks, with or without supervised resistance training.
  Interventions: Drug: Clenbuterol
- Placebo (Placebo Comparator): Participants are randomized to daily ingestion of placebo for a period of 8 weeks, with or without supervised resistance training.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clenbuterol — Participants ingest 80 micrograms clenbuterol daily during the initial 8-week period. This period is followed by a washout of 16 weeks with no drug and resistance training. Thereafter, an 8-week period with supervised resistance training is commenced, with no drug.
  Arms: Clenbuterol
Drug: Placebo — Participants ingest placebo tablets daily during the initial 8-week period. This period is followed by a washout of 16 weeks with no drug and resistance training. Thereafter, an 8-week period with supervised resistance training is commenced, with no drug.
  Arms: Placebo

SUMMARY:
The purpose of the project is investigate muscle memory and underlying mechanisms in humans following resistance training and use of the anabolic substance clenbuterol.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* BMI of <26 and normal ECG and blood pressure

Exclusion Criteria:

* Smoking
* Chronic disease,
* Use of prescription medication
* Pain due to current or previous musculoskeletal injury
* Resistance training more than once per week in the 12 months leading up to the intervention
* Current or previous use of prohibited anabolic substances

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Fiber cross-sectional area | The change in fiber cross-sectional is assessed at baseline, 8, 24 and 32 weeks
  Immunohistochemistry to determine fiber cross-sectional area
Myonuclei | The change in myonuclei is assessed at baseline, 8, 24 and 32 weeks
  Immunohistochemistry to determine number of myonuclei
Skeletal muscle proteome | The change in the muscle proteome is assessed at baseline, 8, 24 and 32 weeks
  Pathway enrichment analysis of the muscle proteome using mass-spectrometry based proteomics

SECONDARY OUTCOMES:
Lean mass | The change in lean mass is assessed at baseline, 8, 24 and 32 weeks
  Lean mass assessed by dual X-ray absorptiometry (DXA)
Isometric muscle strength | The change in maximal voluntary isometric contraction is assessed at baseline, 8, 24 and 32 weeks
  Maximal voluntary isometric contraction of m. quadriceps
Dynamic muscle strength | The change in 1-repetition maximum is assessed at baseline, 8, 24 and 32 weeks
  1-repetition maximum
Sprint performance | The change in sprint performance is assessed at baseline, 8, 24 and 32 weeks
  Work performed (W) during a sprint on a bicycle ergometer
Satellite cells | The change in satellite cells is assessed at baseline, 8, 24 and 32 weeks
  Immunohistochemistry to determine number of satellite cells

CONTACTS AND LOCATIONS:
Locations (1):
- August Krogh Building, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided